CLINICAL TRIAL: NCT02901444
Title: Observational Study on Changing the Quality of Life in Daily Life Activities After Clinical Approach Positioning the Wheelchair
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2015/EV-01
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-09

CONDITIONS: Mobility Limitation; Wheelchairs
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Stemming from the common practice of attribution of the technical helps in the posture in Canada, the multidisciplinary approach of positioning develops in France for more than 10 years old.

To date, no observatory study was led to estimate the impact of such consultation in daily activities, an essential objective conditioning the observance and the acceptance of assistive devices. This study wants to estimate the impact through modification of WHOM scale.

ELIGIBILITY:
Inclusion Criteria:

* persons which are in wheelchair since more than 6 months,
* no recent medical decompensation (<1 mois)

Exclusion Criteria:

* recent medical decompensation

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Personns which are in wheelchair since more than 6 months
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-03; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
WHOM scale (before consultation, after consultation) | 1 month